CLINICAL TRIAL: NCT00710567
Title: Evaluation of the Safety and Effectiveness of the DuraHeart™ Left Ventricular Assist System in Patients Awaiting Transplantation
Brief Title: Evaluation of the Safety and Effectiveness of the DuraHeart™ LVAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Terumo Heart Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DH003
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; LVAS; LVAD; Rotary Pump
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Historical Data (Other): DuraHeart Patients will be implanted with a DuraHeart Left Ventricular Assist System (LVAS) as a "bridge to transplant" until a suitable heart can be found as a replacement. Parameters collected will be compared to a performance goal based on historical data for congestive heart failure patients
  Interventions: Device: DuraHeart Left Ventricular Assist System (LVAS)

INTERVENTIONS:
Device: DuraHeart Left Ventricular Assist System (LVAS) — The DuraHeart LVAS is implanted in using open heart surgery
  Other Names: LVAD

SUMMARY:
Specific Aims The aims of this trial are to evaluate the safety and effectiveness of the DuraHeart™ LVAS in patients with advanced heart failure who require LVAS support as a bridge to cardiac transplantation.

Study Population The patient population for this trial consists of patients with end stage heart failure awaiting cardiac transplantation. Patients must be listed for transplant with UNOS with status 1A or 1B. All patients who meet the eligibility criteria may be included in the study regardless of gender, race or ethnicity.

Study Design This is a multi-center, prospective, single arm study in which the lower one-sided confidence interval exceeds the performance goal. Enrollment is expected to occur within an 18-month time period at up to 40 centers. All patients will be followed for all endpoints for 6 months while on DuraHeart™ LVAS support, or until cardiac transplantation or death, whichever occurs first. For those patients who remain on support after 180 days, survival and device reliability data will continue to be collected on a regular basis. If patients are transplanted, survival at day 30 post cardiac transplantation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

The following are general criteria; more specific conditions are included in the study protocol:

1. Approved for cardiac transplantation
2. Listed with UNOS on the Status 1 list
3. Patient for whom LVAS implantation is planned as a clinically indicated bridge to cardiac transplantation

Exclusion Criteria:

The following are general criteria; more specific conditions are included in the study protocol:

1. Contraindication to the administration of warfarin or anti-platelet agents
2. Primary coagulopathy or platelet disorder
3. Acute myocardial infarction within 48 hours prior to enrollment
4. Anticipated need for RVAD support or ECMO at the time of LVAS implantation
5. Prior cardiac transplantation, left ventricular reduction surgery, cardiomyoplasty, passive restraint device (i.e., CorCapTM Cardiac Support Device) or surgically implanted left ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Survival to cardiac transplantation or to 180 days post implantation and listed for cardiac transplantation in categories UNOS 1A or 1B. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Francis D. Pagani, M.D., Ph.D., Principal Investigator — University of Michigan; Yoshifumi Naka, M.D., Ph.D., Principal Investigator — Columbia University; David S Feldman, MD, Principal Investigator — Minneapolis Heart Institute
Locations (26):
- United States (25):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - St. Vincent Hospital, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Minneapoils Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Newark Beth Israel, Newark, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Penn State University, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical City, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No